CLINICAL TRIAL: NCT05913232
Title: A Phase 2b Randomized, Double-masked, Active-controlled, Dose-response Study of the Safety and Efficacy of H-1337 in Subjects With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension
Brief Title: Study of Safety and Efficacy of H-1337 in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: D. Western Therapeutics Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H1337-CS202
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Glaucoma Open-Angle Primary; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- H-1337 0.6% Ophthalmic Solution b.i.d. (Experimental): One drop H-1337 twice daily in the study eye for 28 days
  Interventions: Drug: H-1337 0.6%
- H-1337 1.0% Ophthalmic Solution b.i.d. (Experimental): One drop H-1337 twice daily in the study eye for 28 days
  Interventions: Drug: H-1337 1.0%
- H-1337 1.0% Ophthalmic Solution q.a.m. and H-1337 Placebo q.p.m. (Experimental): One drop H-1337 every morning and matching placebo every evening in the study eye for 28 days
  Interventions: Drug: H-1337 1.0%; Drug: H-1337 Placebo
- Timolol 0.5% Ophthalmic Solution b.i.d. (Active Comparator): One drop Timolol twice daily in the study eye for 28 days
  Interventions: Drug: Timolol 0.5%

INTERVENTIONS:
Drug: H-1337 0.6% — ophthalmic solution
  Arms: H-1337 0.6% Ophthalmic Solution b.i.d.
Drug: H-1337 1.0% — ophthalmic solution
  Arms: H-1337 1.0% Ophthalmic Solution b.i.d.; H-1337 1.0% Ophthalmic Solution q.a.m. and H-1337 Placebo q.p.m.
Drug: H-1337 Placebo — ophthalmic solution
  Arms: H-1337 1.0% Ophthalmic Solution q.a.m. and H-1337 Placebo q.p.m.
Drug: Timolol 0.5% — ophthalmic solution
  Arms: Timolol 0.5% Ophthalmic Solution b.i.d.

SUMMARY:
The trial will evaluate the safety and efficacy of 3 dose regimens of H-1337 [0.6% twice daily (b.i.d.), 1.0% b.i.d. and 1.0% once in the morning (q.a.m.), and timolol maleate (0.5%, b.i.d.) in both eyes for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral primary open angle glaucoma or ocular hypertension

Exclusion Criteria:

* Closed or very narrow angles (Grades 0-1) or those the investigator judges as occludable and/or with evidence of peripheral anterior synechiae >/= 180 degrees by gonioscopy within 6 months prior to screening visit in either eye

Note: Other inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: El-Roy Dixon, MD, Principal Investigator — Dixon Eye Care
Locations (9):
- United States (9):
  - Global Research Management, Glendale, California
  - Skyline Vision Clinic and Laser Center, Colorado Springs, Colorado
  - Central Florida Eye Associates, Lakeland, Florida
  - Shettle Eye Research, Inc., Largo, Florida
  - Dixon Eye Care, Albany, Georgia
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - University Eye Specialists, Maryville, Tennessee
  - Vistar Eye Center, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A 49-day screening period (screening visit plus washout period) occurred prior to randomization and the treatment period.
Period: Overall Study
Arm/Group | H-1337 0.6% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution q.a.m. and H-1337 Placebo q.p.m. | Timolol 0.5% Ophthalmic Solution b.i.d.
Started | 51 | 51 | 50 | 49
Completed | 51 | 49 | 49 | 48
Not Completed | 0 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H-1337 0.6% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution q.a.m. and H-1337 Placebo q.p.m. | Timolol 0.5% Ophthalmic Solution b.i.d. | Total
Number analyzed (Participants) | 51 | 51 | 50 | 49 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 21 | 19 | 27 | 92
  >=65 years | 26 | 30 | 31 | 22 | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 26 | 19 | 97
  Male | 25 | 25 | 24 | 30 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 7 | 5 | 29
  Not Hispanic or Latino | 43 | 42 | 43 | 44 | 172
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 14 | 13 | 15 | 17 | 59
  White | 36 | 36 | 35 | 32 | 139
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Iris Color [Count of Participants; unit: Participants]
  Brown | 30 | 28 | 30 | 34 | 122
  Blue | 10 | 9 | 13 | 9 | 41
  Green | 2 | 4 | 1 | 2 | 9
  Hazel | 9 | 9 | 3 | 3 | 24
  Other | 0 | 1 | 3 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Assessed by Change in Intraocular Pressure
Description: Mean change in intraocular pressure from baseline on Day 28 compared to timolol
Time Frame: Day 28
Population: Intent-to-Treat (ITT) is defined as all randomized subjects.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: study eyes
Arm/Group | H-1337 0.6% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution q.a.m. and H-1337 Placebo q.p.m. | Timolol 0.5% Ophthalmic Solution b.i.d.
Number analyzed (Participants) | 51 | 51 | 50 | 49
Number analyzed (study eyes) | 51 | 51 | 50 | 49
mmHg
  Day 28: Pre T0, change from baseline (mmHg): number analyzed (Participants) | 51 | 50 | 49 | 48
  Day 28: Pre T0, change from baseline (mmHg): number analyzed (study eyes) | 51 | 50 | 49 | 48
  Day 28: Pre T0, change from baseline (mmHg) | -6.3 (3.27) | -6.3 (3.15) | -5.9 (3.45) | -7.0 (3.26)
  Day 28: T0 + 2h, change from baseline (mmHg): number analyzed (Participants) | 51 | 49 | 49 | 48
  Day 28: T0 + 2h, change from baseline (mmHg): number analyzed (study eyes) | 51 | 49 | 49 | 48
  Day 28: T0 + 2h, change from baseline (mmHg) | -7.3 (3.07) | -7.2 (3.14) | -6.5 (3.67) | -6.3 (3.83)
  Day 28: T0 + 4h, change from baseline (mmHg): number analyzed (Participants) | 51 | 49 | 49 | 48
  Day 28: T0 + 4h, change from baseline (mmHg): number analyzed (study eyes) | 51 | 49 | 49 | 48
  Day 28: T0 + 4h, change from baseline (mmHg) | -7.5 (3.28) | -7.3 (3.24) | -6.8 (3.48) | -5.3 (3.53)
  Day 28: T0 + 8h, change from baseline (mmHg): number analyzed (Participants) | 51 | 49 | 49 | 48
  Day 28: T0 + 8h, change from baseline (mmHg): number analyzed (study eyes) | 51 | 49 | 49 | 48
  Day 28: T0 + 8h, change from baseline (mmHg) | -6.8 (3.67) | -6.5 (3.50) | -6.1 (3.12) | -5.3 (3.21)
  Day 28: T0 + 12h, change from baseline (mmHg): number analyzed (Participants) | 46 | 45 | 45 | 45
  Day 28: T0 + 12h, change from baseline (mmHg): number analyzed (study eyes) | 46 | 45 | 45 | 45
  Day 28: T0 + 12h, change from baseline (mmHg) | -5.6 (3.82) | -5.3 (3.37) | -5.5 (3.44) | -4.9 (3.35)
  Day 28: 8-hour diurnal, change from baseline (mmHg): number analyzed (Participants) | 51 | 49 | 49 | 48
  Day 28: 8-hour diurnal, change from baseline (mmHg): number analyzed (study eyes) | 51 | 49 | 49 | 48
  Day 28: 8-hour diurnal, change from baseline (mmHg) | -7.2 (3.04) | -7.0 (2.90) | -6.4 (3.14) | -5.6 (3.16)
  Day 28: 12-hour diurnal, change from baseline (mmHg): number analyzed (Participants) | 51 | 49 | 49 | 48
  Day 28: 12-hour diurnal, change from baseline (mmHg): number analyzed (study eyes) | 51 | 49 | 49 | 48
  Day 28: 12-hour diurnal, change from baseline (mmHg) | -6.8 (3.02) | -6.6 (2.76) | -6.2 (3.11) | -5.4 (2.99)

2. Secondary Outcome: Efficacy as Assessed by Intraocular Pressure
Description: Percentage of subjects reaching target intraocular pressure (≤18 mmHg) at each time point
Time Frame: Day 0, Day 1, Day 7, Day 14, and Day 28
Population: Intent-to-Treat (ITT) is defined as all randomized subjects.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Units Other Than Participants: study eyes
Arm/Group | H-1337 0.6% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution q.a.m. and H-1337 Placebo q.p.m. | Timolol 0.5% Ophthalmic Solution b.i.d.
Number analyzed (Participants) | 51 | 51 | 50 | 49
Number analyzed (study eyes) | 51 | 51 | 50 | 49
percentage of subjects
  Day 0: Pre T0 | 0.0 [0.0 to 7.0] | 2.0 [0.0 to 10.4] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 7.3]
  Day 0: T0 + 2h | 0.0 [0.0 to 7.0] | 3.9 [0.5 to 13.5] | 4.0 [0.5 to 13.7] | 2.0 [0.1 to 10.9]
  Day 0: T0 + 4h | 2.0 [0.0 to 10.4] | 2.0 [0.0 to 10.4] | 2.0 [0.1 to 10.6] | 2.0 [0.1 to 10.9]
  Day 0: T0 + 8h | 5.9 [1.2 to 16.2] | 3.9 [0.5 to 13.5] | 6.0 [1.3 to 16.5] | 6.1 [1.3 to 16.9]
  Day 0: T0 + 12h | 10.9 [3.6 to 23.6] | 10.9 [3.6 to 23.6] | 15.2 [6.3 to 28.9] | 13.3 [5.1 to 26.8]
  Day 0: 12-hour diurnal | 2.0 [0.0 to 10.4] | 2.0 [0.0 to 10.4] | 2.0 [0.1 to 10.6] | 2.0 [0.1 to 10.9]
  Day 0: 8-hour diurnal | 0.0 [0.0 to 7.0] | 2.0 [0.0 to 10.4] | 2.0 [0.1 to 10.6] | 2.0 [0.1 to 10.9]
  Day 1: Pre T0 | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 7.3]
  Day 1: T0 + 2h | 31.4 [19.1 to 45.9] | 35.3 [22.4 to 49.9] | 28.0 [16.2 to 42.5] | 46.9 [32.5 to 61.7]
  Day 1: T0 + 4h | 51.0 [36.6 to 65.2] | 58.8 [44.2 to 72.4] | 70.0 [55.4 to 82.1] | 63.3 [48.3 to 76.6]
  Day 1: T0 + 8h | 60.8 [46.1 to 74.2] | 68.6 [54.1 to 80.9] | 74.0 [59.7 to 85.4] | 61.2 [46.2 to 74.8]
  Day 1: T0 + 12h | 67.4 [52.0 to 80.5] | 72.3 [57.4 to 84.4] | 84.4 [70.5 to 93.5] | 76.1 [61.2 to 87.4]
  Day 1: 12-hour diurnal | 54.9 [40.3 to 68.9] | 54.9 [40.3 to 68.9] | 52.0 [37.4 to 66.3] | 53.1 [38.3 to 67.5]
  Day 1: 8-hour diurnal | 47.1 [32.9 to 61.5] | 51.0 [36.6 to 65.2] | 52.0 [37.4 to 66.3] | 53.1 [38.3 to 67.5]
  Day 7: Pre T0 | 37.3 [24.1 to 51.9] | 30.0 [17.9 to 44.6] | 20.4 [10.2 to 34.3] | 44.9 [30.7 to 59.8]
  Day 14: Pre T0 | 41.2 [27.6 to 55.8] | 36.0 [22.9 to 50.8] | 26.5 [14.9 to 41.1] | 47.9 [33.3 to 62.8]
  Day 28: Pre T0 | 31.4 [19.1 to 45.9] | 40.0 [26.4 to 54.8] | 34.7 [21.7 to 49.6] | 52.1 [37.2 to 66.7]
  Day 28: T0 + 2h | 66.7 [52.1 to 79.2] | 63.3 [48.3 to 76.6] | 55.1 [40.2 to 69.3] | 58.3 [43.2 to 72.4]
  Day 28: T0 + 4h | 74.5 [60.4 to 85.7] | 81.6 [68.0 to 91.2] | 79.6 [65.7 to 89.8] | 52.1 [37.2 to 66.7]
  Day 28: T0 + 8h | 68.6 [54.1 to 80.9] | 77.6 [63.4 to 88.2] | 67.3 [52.5 to 80.1] | 62.5 [47.4 to 76.0]
  Day 28: T0 + 12h | 67.4 [52.0 to 80.5] | 68.9 [53.4 to 81.8] | 71.1 [55.7 to 83.6] | 64.4 [48.8 to 78.1]
  Day 28: 12-hour diurnal | 58.8 [44.2 to 72.4] | 63.3 [48.3 to 76.6] | 65.3 [50.4 to 78.3] | 54.2 [39.2 to 68.6]
  Day 28: 8-hour diurnal | 64.7 [50.1 to 77.6] | 67.3 [52.5 to 80.1] | 65.3 [50.4 to 78.3] | 50.0 [35.2 to 64.8]

3. Secondary Outcome: Safety as Assessed by Adverse Event Reporting
Description: Percentage of participants with ocular and systemic adverse events
Time Frame: Screening through Day 28
Population: Safety population is defined as all randomized subjects who received at least one dose of investigational product.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | H-1337 0.6% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution q.a.m. and H-1337 Placebo q.p.m. | Timolol 0.5% Ophthalmic Solution b.i.d.
Number analyzed (Participants) | 51 | 51 | 50 | 49
percentage of subjects
  Ocular Treatment-Emergent Adverse Events | 43.1 [29.3 to 57.8] | 60.8 [46.1 to 74.2] | 64.0 [49.2 to 77.1] | 18.4 [8.8 to 32.0]
  Systemic Treatment-Emergent Adverse Events | 3.9 [0.5 to 13.5] | 7.8 [2.2 to 18.9] | 4.0 [0.5 to 13.7] | 2.0 [0.1 to 10.9]

ADVERSE EVENTS:
Time Frame: 28 days
Description: Treatment-emergent adverse events (TEAE) are defined as AEs starting on or after the first dose of IP. A pre-existing event that worsens in severity after receiving the first dose of IP is treated as a new TEAE with date of onset set to the date of the increased severity.
  An ocular event is an event where the site of the event is reported as both eyes (OU), right eye (OD) or left eye (OS).
Arm/Group | H-1337 0.6% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution b.i.d. | H-1337 1.0% Ophthalmic Solution q.a.m. and H-1337 Placebo q.p.m. | Timolol 0.5% Ophthalmic Solution b.i.d.
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51 | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 19/51 | 28/51 | 29/50 | 8/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H-1337 0.6% Ophthalmic Solution b.i.d. (N=51) | H-1337 1.0% Ophthalmic Solution b.i.d. (N=51) | H-1337 1.0% Ophthalmic Solution q.a.m. and H-1337 Placebo q.p.m. (N=50) | Timolol 0.5% Ophthalmic Solution b.i.d. (N=49)
Conjunctival hyperaemia (Eye disorders) | 16 (25) | 19 (30) | 26 (44) | 5 (6) — Hyperemia was coded as conjunctival hyperemia if it was specifically indicated as occurring in the conjunctiva; all other cases of hyperemia were coded as ocular hyperemia.
Instillation site irritation (General disorders) | 7 (7) | 11 (11) | 7 (7) | 3 (3)

LIMITATIONS AND CAVEATS:
No significant limitations or caveats were reported for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT05913232/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT05913232/SAP_001.pdf